CLINICAL TRIAL: NCT02233959
Title: Palatability of a Novel Oral Formulation of Prednsione
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: Orbis (Other)
Responsible Party: Principal Investigator, Greg Kearns, Senior Vice President and Chief Research Officer, Arkansas Children's Hospital Research Institute
Other Study IDs: Orbis Palatability
Record Dates: First submitted 2014-09-03; First posted 2014-09-09 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Palatability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Adults

SUMMARY:
Prednisone solution USP (5mg/5mL), is the most commonly prescribed formulation of prednisone to pediatric and adult patients. The rationale for this study is that palatability is the most important determinant of pediatric patient compliance, and therefore, it is critical that the Orbis formulation be perceived as significantly more palatable compared to today's commercially available products in order to warrant further development of the TP.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 32 years, male and female who are healthy at the time of study
* can demonstrate holding 10 mL of apple juice in mouth for 5 seconds without swallowing and then expectorate contents into a cup
* demonstrate ability to complete study questionnaire

Exclusion Criteria:

* history of smoking or using any tobacco products
* previous history of taste disturbance
* any condition or dietary habit known to interfere with the sense of smell and taste
* any structural or functional abnormality of the upper gastrointestinal tract
* ingestion of any medication or nutritional supplement (with exception of acetaminophen tablets or capsules) in a 48 hour period prior to study
* history of any significant illness within the two weeks prior to study
* history of autonomic dysfunction, bronchospastic disease or atopic allergy
* known hypersensitivity (ie., allergic reaction) to any drug, food coloring agent or artificial sweetener
* any history of participating in a clinical trial of a drug or device within a 30 day period from the time of study
* brushing of the teeth, usage of mouthwash, and or oral ingestion of any substance within two hours of receipt of the initial test article and
* inability to speak and/or read English at a grade 10 level

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 24 healthy young adults (12 males and 12 females), ranging in age from 18 to 32 years of age comprised of a convenience sample who meet study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Palatability of a new oral formulation of prednisone | Immediately
  We will create optimized shelf-stable prednisone microcapsules designed for complete taste-masking followed by immediate release in the stomach. Release characteristics of the TP will be compared to a pharmaceutical grade formulation of prednisone. Milestone: Microencapsulated prednisone that: (i) shows less than 10% coefficient of variance (CV) in the in vitro release profile between fresh and 4-week, 40°C stability-exposed samples while maintaining (ii) maximum of 5% total drug release during the initial 2 minutes and (iii) >90% release within 30 minutes.
  N.B. This Specific Aim will be accomplished in the laboratories of Orbis Biosciences, Inc. Upon meeting all milestones associated with this SA, Orbis Biosciences will produce, in accordance with Good Laboratory and Manufacturing Principles, a single batch of TP suitable for use in accomplish SA2.

SECONDARY OUTCOMES:
Evaluation of the TP for the organoleptic properties of taste, mouth-feel and aroma in healthy adults compared to the reference product (RP). | Immediately
  We will use a randomized cross-over design and a 9-Point Hedonic bipolar scale of scoring to compare the product appearance, smell, taste, mouth feel and after taste for three treatment groups: (i) Orbis's prednisone-loaded microcapsules (TP), developed in SA1, (ii) TP placebo microcapsules (i.e., delivery system not containing any active pharmaceutical ingredient or API), and (iii) the RP (Prednisone oral liquid, USP). We will suspend the microcapsules in a non-flavored suspension medium immediately before administration to healthy adults. The hypothesis associated with this SA is that microencapsulated prednisone (TP) will demonstrate significant improvement in organoleptic properties as compared to the RP.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Kearns, Pharm D. PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided